CLINICAL TRIAL: NCT04739917
Title: Safety and Protective Efficacy of a Synthetic Vaccine Derived From the CS Protein of Plasmodium Vivax: a Double-blind, Placebo-controlled, Randomized Clinical Trial in naïve and Pre-immune Colombian Volunteers
Brief Title: Efficacy of a Synthetic Vaccine Derived From Plasmodium Vivax Circumsporozoite Protein (PvCS) in naïve and Semi-immune Volunteers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Malaria Vaccine and Drug Development Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MVDC-2021-001
Record Dates: First submitted 2021-01-25; First posted 2021-02-05 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Malaria, Vivax
Keywords: Malaria; Vaccine; Vivax
MeSH Terms: conditions — Malaria, Vivax; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm N Vaccine (Experimental): 30 malaria-naïve subjects from non-endemic areas of Cali, Colombia.
  Interventions: Biological: Vaccine PvCS N+C+R 150 mcg
- Arm N Placebo (Placebo Comparator): 30 malaria-naïve subjects from non-endemic areas of Cali, Colombia.
  Interventions: Other: Placebo SSN Montanide ISA-51 1 mL
- Arm S Vaccine (Experimental): 30 semi-immune subjects from malaria endemic areas of Chocó, Colombia.
  Interventions: Biological: Vaccine PvCS N+C+R 150 mcg
- Arm S Placebo (Placebo Comparator): 30 semi-immune subjects from malaria endemic areas of Chocó, Colombia.
  Interventions: Other: Placebo SSN Montanide ISA-51 1 mL

INTERVENTIONS:
Biological: Vaccine PvCS N+C+R 150 mcg — Vaccine PvCS N+C+R 150 mcg (Montanide ISA-51), freeze dried powder.
  Arms: Arm N Vaccine; Arm S Vaccine
Other: Placebo SSN Montanide ISA-51 1 mL — SSN Montanide ISA-51 1 mL
  Arms: Arm N Placebo; Arm S Placebo

SUMMARY:
This is a randomized, double-blind, controlled, which seeks to compare two groups of volunteers (naive and previously exposed to malaria) vaccinated with three doses of a synthetic derivative of the CS protein of Plasmodium vivax to determine their protective efficacy.

Then volunteers will be subject to an infectious challenge (Controlled Human Malaria Infection) to assess the infectivity of gametocytes in the blood early stage of P. vivax in Anopheles albimanus mosquitoes.

DETAILED DESCRIPTION:
This study is a prospective controlled, blinded clinical trial, designed to establish the protective efficacy induced by the vaccine PvCSP between human volunteers with and without history of malaria. Volunteers will be recruited in Cali, Colombia and Quibdó, Colombia.

Study subjects: This study will require the involvement of two types of volunteers, parasite donors and volunteers for immunization

Parasite donors: 5-15 P. vivax-infected patients who will serve as parasites donors for experimental infection of mosquitoes, who will be enrolled in the endemic area.

Volunteers for immunization: Two other groups of volunteers will be immunized with the PvCSP vaccine. A group of 60 people without previous exposure to malaria (naïve) and another 60 people with a history of previous malaria infection (pre-immune).

Methodology Recruitment of infected patients: Parasite donors will be recruited among P. vivax infected patients attending a diagnostic center in the endemic area.

Infection of mosquito's blood from donors will be used to feed three-day-old mosquitoes by artificial membrane feeding technique. At day 7, a sample of mosquitoes will be examined to determine the level of infection by dissection of the mosquito's gut. On day 14, a small number of mosquitoes with a good degree of infectivity will be used to infect challenged volunteers.

Recruitment of pre-immune and naive volunteers: Volunteers for the immunization stage will be recruited both in the city of Cali (Colombia), non-endemic region, and in Quibdó (Colombia), a malaria endemic region, through various activities such as conferences, meetings and other strategies previously approved by the IRB, like posters, radio advertising flyers and social media.

Immunization: Volunteers will be immunized with the vaccine (n=60) or placebo (n=60).

Follow-up of volunteers will be performed under medical vigilance during the first hour following the immunization to detect any adverse reaction. After the first hour period a medical exam will be made. Eight hours after immunization, each volunteer will be contacted via telephone to assess physical condition. Any adverse event (AE) will be registered.

Subsequent follow up will be made on the day next to immunization and 1 or 2 weeks before the next immunization by a new clinical evaluation and AE report. Volunteers will be instructed to contact the research staff at any moment.

Infection of volunteers immunized volunteers will be challenged on day ~150 of the study, 1 month after the third immunization by the bite of 2-4 infected mosquito. A "feeding cage" will be placed on the forearm of a volunteer for 10 minutes, allowing that the feeding window, which will be covered by a mesh surface be placed against the volunteer's skin.

Volunteers will be instructed about the signs and symptoms of malaria and they will have a daily telephone contact during the first 6 days.

Between days 7 and 23 the volunteers will be asked to go to the Clinical Trials Unit daily to establish the presence or absence of disease through thick blood smear and samples will be collected for retrospective real time PCR P. vivax.

From day 23 until day 31, volunteers will receive physical and laboratory evaluation every other day and will have daily telephone contact.

Once the patients present signs and symptoms of the disease curative treatment will be immediately provided, and 15 ml of blood will be drawn, which will be used for immune response assessment.

If the volunteers do not develop the disease during the follow-up period, on day 31 they will be given antimalarial treatment.

Treatment Volunteers will be treated with antimalarial drugs approved by the Colombian Ministry of Social Health: chloroquine (three (3) doses: 600 mg initially, followed by 450 mg at 24, and 48 hours), associated with primaquine (30mg/day) for 14 days. All the volunteers will be asked to return two weeks after starting treatment for a thick blood smear test to ensure cure of malaria.

ELIGIBILITY:
Inclusion Criteria:

Naïve group:

1. Non-pregnant, healthy men and women between 18-45 years old.
2. Freely and voluntarily sign an IC, accompanied by two witnesses who must also sign.
3. Absence history of malaria infection.
4. To have negative serology for the PvCS protein by the ELISA test.
5. For women, not be pregnant.
6. Use of an adequate contraceptive method from the beginning until the contraceptive restriction is lifted by a study doctor, at the end of the study.
7. To accept not to travel to areas considered as endemic for malaria from the infectious challenge period and to the end of its follow-up (1 month).
8. Be reachable by phone throughout the study period.
9. To be Duffy positive (Fy +).
10. Have Hemoglobin (Hb) levels> 11 g / dl.
11. Be willing to participate during the period in which the study will take place.
12. Not be participating in another clinical study.
13. Be affiliated with the general health social security system of Colombia, in any of its regimes (subsidized or contributory)

Semi-immune group:

1. Non-pregnant, healthy men and women between 18-45 years old,
2. Freely and voluntarily sign an informed consent, accompanied by two witnesses who will also sign.
3. Have a history of malaria infection (s) and positive serological tests (ELISA) for P. vivax.
4. For women, not be pregnant or nursing.
5. For women, use of adequate contraception from inception until the contraceptive restriction is lifted by a study physician.
6. Be a permanent resident of the municipality of Quibdó during the study.
7. Be reachable by phone throughout the study period.
8. Availability to participate during the period in which the study will take place.
9. Be affiliated with the general health social security system of Colombia, in any of its regimes (subsidized or contributory)

Exclusion Criteria:

Naïve group:

1. Glucose 6 phosphate dehydrogenase deficiency (G-6-P-D).
2. Present any hemoglobinopathy (eg HbS).
3. Personal history of allergies to medications or insect bites.
4. Have received vaccination against malaria.
5. Clinical or laboratory abnormalities determined by the investigator (s).
6. IFAT> 1:20 for P. vivax in screening tests.
7. Have lived in a malaria-endemic region during the 12 months before the study.
8. Clinical or laboratory evidence of systemic disease, including kidney, liver, cardiovascular, pulmonary, psychiatric, or other diseases that may negatively impact and alter study results.
9. Evidence of active hepatitis B or Hepatitis C infection
10. Evidence of active HIV infection.
11. History of transfusion of any blood product in the 6 (six) months before the study.
12. Plan to have surgery from the recruitment period to the end of the post-challenge follow-ups.
13. Presence or history of autoimmune disease (lupus, rheumatoid arthritis, thyroiditis, or other).
14. Splenectomized volunteers.
15. Volunteers in treatment with drugs with activity on the immune system (steroids, immunosuppressive agents, or immunomodulators).
16. History of alcoholism or drug abuse defined as a habit that interferes with the normal social functioning of the individual.
17. Any condition that may interfere with the ability to provide a free and voluntary IC.
18. Not being affiliated with the general health social security system of Colombia, in any of its regimes (subsidized or contributory)

Semi-immune group:

1. IFAT negative (<1:20) for P. vivax in screening tests.
2. The other criteria used in the case of naïve volunteers, except the antecedent of having lived in the endemic area.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of first case of P. vivax malaria after CHMI and meeting the primary case definition. | Assessed over average of 16-18 days post CHMI (range 7 to 60 days)
  The first case of malaria meeting the primary case definition will be defined as the first or only episodes with the presence of Plasmodium vivax parasitemia ≥ 0.1% by thick blood smear and malaria qPCR.

SECONDARY OUTCOMES:
Concentration of specific anti-PvCS IgG antibodies IgG (isotypes) against the different functional fragments of the Pv-CS protein. | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Concentration of specific anti-PvCS IgG antibodies IgG (isotypes) against the different functional fragments of the Pv-CS protein (Amino, Central Repeat and Carboxilo terminal). Expressed both as antibody titers and Reactive Indices (RI) measured by in enzyme-linked immunosorbent assay (ELISA) and Immunofluorescence Test (IFAT). Antibody titers by IFAT are determine as the reciprocal of the end-points dilution showing a positive fluorescence.
  Concentrations will be presented as geometric mean concentrations (GMCs).
Specific cytokine induction | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Specific cytokine induction will be measured by IFN- γ, TNF-α, IL-2; IL- 4, IL-6, IL-10
T-cell response measurement - Flow cytometry | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  In vitro proliferation of CD3+ T-cells (CD4+ and CD8+) and intracellular production of cytokines IFN-gamma, TNF-a, IL-12 by flow cytometry. Result will be expressed as percentages.
T-cell response measurement - ELIspot | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Production of IFN-gamma and IL-10 in total PBMC stimulated with the different antigens and / or synthetic peptides by ELIspot assay. Results expressed as the mean number of IFN-γ spot-forming cells (sfc) per 106 Peripheral Blood Mononuclear Cells.
T-cell response measurement - Bioplex | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Multiplex cytokines profile (Th1/Th2/Treg) in sera by bioplex. Cytokine concentrations were calculated from the standard curve using seven-parameter curve fitting software and the results were expressed in pg/mL. The limit of detection for the assay was 10 pg/mL for all cytokines. Results will be expressed as percentages.
Characterization of T lymphocytes | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Phenotyping and profiles of memory T lymphocytes will be done in PBMCs using specific panels of markers by flow cytometry. The frequency of cells as a biomarker post CHMI infection will be performed. Cells will be stained by using different antibody cocktails targeting specific cell populations. Cells acquisition will be done on a 4-laser BD flow cytometer and gating analysis with FlowJo software version 10.4.2. Results will be expressed as percentages.
Characterization of B lymphocytes. | Days 0, 30, 60, 90, 120, 180, 210 and 240
  Phenotyping and profiles of B lymphocytes will be done in PBMCs using specific panels of markers by flow cytometry. The frequency of cells as a biomarker post CHMI infection will be performed. Cells will be stained by using different antibody cocktails targeting specific cell populations. Cells acquisition will be done on a 4-laser BD flow cytometer and gating analysis with FlowJo software version 10.4.2. Results will be expressed as percentages.
Characterization of monocytes | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Phenotyping and profiles of monocytes will be done in PBMCs using specific panels of markers by flow cytometry. The frequency of cells as a biomarker post CHMI infection will be performed. Cells will be stained by using different antibody cocktails targeting specific cell populations. Cells acquisition will be done on a 4-laser BD flow cytometer and gating analysis with FlowJo software version 10.4.2. Results will be expressed as percentages.
Antibody functionality in vitro through inhibition of sporozoite invasion (ISI) to Hep-G2 cells. | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Antibody functionality will be tested in vitro through essays of inhibition of sporozoite invasion (ISI) to Hep-G2 cells.
Vaccine-induced protection for P. vivax | Thirty days after mosquito bite challenge (Controlled Human Malaria Infection)
  Vaccine-induced protection for P. vivax will be assessed by pre-patent period onset after infected mosquito bites exposure
Multiomics testing (i.e., transcriptomics, genomics) | Days 0, 30, 90, 195 and 225.
  Tthe present study also seeks to evaluate host-related variables, especially those affected by the immune status prior to vaccination (naïve vs pre-immune participants).
  To accomplish this, transcriptomics and genomics tests will be undertaken on days 0, 30, 195 and, 225.
Safety - Number of Subjects With Any and Grade 3 Solicited Local Symptoms | During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
  Assessed solicited local symptoms will be pain and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 swelling = swelling spreading beyond 20 millimeters (mm) of injection site.
Safety - Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms | During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
  Assessed solicited general symptoms will be drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite.
  Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity.
  Grade 3 fever = fever higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Safety - Number of Subjects With Any Unsolicited Adverse Events (AEs) | Within the 30-day (Days 0-29) post-vaccination follow-up period
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Any will be defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Safety - Number of Subjects With Serious Adverse Events (SAEs) | Throughout the study period (Day 0 - Month 14)
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Safety - Number of Subjects With Hemoglobin Values Outside Normal Ranges With Toxicity Grades | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With White Blood Cell (WBC) Values Outside Normal Ranges With Toxicity Grades | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Platelet Values Outside Normal Ranges With Toxicity Grades | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Alanine Aminotransferase (ALT) Values Outside Normal Ranges With Toxicity Grades | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Creatinine Values Outside Normal Ranges With Toxicity Grades | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Bilirubin Values Outside Normal Ranges With Toxicity Grades | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Alkaline phosphatase Values Outside Normal Ranges With Toxicity | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Blood urea nitrogen (BUN) Values Outside Normal Ranges With Toxicity | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Aspartate aminotransferase (AST) Values Outside Normal Ranges With Toxicity | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Prothrombin time (PT)) Values Outside Normal Ranges With Toxicity | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of Subjects With Partial thromboplastin time (PTT) Values Outside Normal Ranges With Toxicity | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Toxicity levels will be measured according to the Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0.
Safety - Number of participants with confirmed pregnancy | Days 0, 30, 60, 90, 120, 180, 210 and 240.
  Number of participants with confirmed pregnancy during the study duration.
Safety - Glucose-6-phosphate dehydrogenase deficiency | Day 0.
  Glucose-6-phosphate dehydrogenase deficiency test will be done during baseline evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Sócrates Herrera, MD, Principal Investigator — Director
Locations (1):
- Malaria Vaccine and Drug Development Center, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Ademolue TW, Awandare GA. Evaluating antidisease immunity to malaria and implications for vaccine design. Immunology. 2018 Apr;153(4):423-434. doi: 10.1111/imm.12877. Epub 2017 Dec 26. PMID 29211303
- [Background] RTS,S Clinical Trials Partnership. Efficacy and safety of the RTS,S/AS01 malaria vaccine during 18 months after vaccination: a phase 3 randomized, controlled trial in children and young infants at 11 African sites. PLoS Med. 2014 Jul 29;11(7):e1001685. doi: 10.1371/journal.pmed.1001685. eCollection 2014 Jul. PMID 25072396
- [Background] Aliprandini E, Tavares J, Panatieri RH, Thiberge S, Yamamoto MM, Silvie O, Ishino T, Yuda M, Dartevelle S, Traincard F, Boscardin SB, Amino R. Cytotoxic anti-circumsporozoite antibodies target malaria sporozoites in the host skin. Nat Microbiol. 2018 Nov;3(11):1224-1233. doi: 10.1038/s41564-018-0254-z. Epub 2018 Oct 22. PMID 30349082
- [Background] Arevalo-Herrera M, Herrera S. Plasmodium vivax malaria vaccine development. Mol Immunol. 2001 Dec;38(6):443-55. doi: 10.1016/s0161-5890(01)00080-3. PMID 11741694
- [Background] Arevalo-Herrera M, Roggero MA, Gonzalez JM, Vergara J, Corradin G, Lopez JA, Herrera S. Mapping and comparison of the B-cell epitopes recognized on the Plasmodium vivax circumsporozoite protein by immune Colombians and immunized Aotus monkeys. Ann Trop Med Parasitol. 1998 Jul;92(5):539-51. PMID 9797827
- [Background] Arevalo-Herrera M, Soto L, Perlaza BL, Cespedes N, Vera O, Lenis AM, Bonelo A, Corradin G, Herrera S. Antibody-mediated and cellular immune responses induced in naive volunteers by vaccination with long synthetic peptides derived from the Plasmodium vivax circumsporozoite protein. Am J Trop Med Hyg. 2011 Feb;84(2 Suppl):35-42. doi: 10.4269/ajtmh.2011.09-0507. PMID 21292876
- [Background] Arevalo-Herrera M, Chitnis C, Herrera S. Current status of Plasmodium vivax vaccine. Hum Vaccin. 2010 Jan;6(1):124-32. doi: 10.4161/hv.6.1.9931. Epub 2010 Jan 26. PMID 20009526
- [Background] Arnot DE, Stewart MJ, Barnwell JW. Antigenic diversity in Thai Plasmodium vivax circumsporozoite proteins. Mol Biochem Parasitol. 1990 Nov;43(1):147-9. doi: 10.1016/0166-6851(90)90140-h. No abstract available. PMID 2290443
- [Background] Arnot DE, Barnwell JW, Tam JP, Nussenzweig V, Nussenzweig RS, Enea V. Circumsporozoite protein of Plasmodium vivax: gene cloning and characterization of the immunodominant epitope. Science. 1985 Nov 15;230(4727):815-8. doi: 10.1126/science.2414847.
- [Background] Barnwell JW, Galinski MR. Plasmodium vivax: a glimpse into the unique and shared biology of the merozoite. Ann Trop Med Parasitol. 1995 Apr;89(2):113-20. doi: 10.1080/00034983.1995.11812941. PMID 7605120
- [Background] Barnwell JW, Galinski MR, DeSimone SG, Perler F, Ingravallo P. Plasmodium vivax, P. cynomolgi, and P. knowlesi: identification of homologue proteins associated with the surface of merozoites. Exp Parasitol. 1999 Mar;91(3):238-49. doi: 10.1006/expr.1998.4372. PMID 10072326
- [Background] Bermudez M, Moreno-Perez DA, Arevalo-Pinzon G, Curtidor H, Patarroyo MA. Plasmodium vivax in vitro continuous culture: the spoke in the wheel. Malar J. 2018 Aug 20;17(1):301. doi: 10.1186/s12936-018-2456-5. PMID 30126427
- [Background] Burkot TR, Wirtz RA, Paru R, Garner P, Alpers MP. The population dynamics in mosquitoes and humans of two Plasmodium vivax polymorphs distinguished by different circumsporozoite protein repeat regions. Am J Trop Med Hyg. 1992 Dec;47(6):778-86. doi: 10.4269/ajtmh.1992.47.778. PMID 1471735
- [Background] Cattani JA, Tulloch JL, Vrbova H, Jolley D, Gibson FD, Moir JS, Heywood PF, Alpers MP, Stevenson A, Clancy R. The epidemiology of malaria in a population surrounding Madang, Papua New Guinea. Am J Trop Med Hyg. 1986 Jan;35(1):3-15. doi: 10.4269/ajtmh.1986.35.3. PMID 3511748
- [Background] Cerami C, Frevert U, Sinnis P, Takacs B, Clavijo P, Santos MJ, Nussenzweig V. The basolateral domain of the hepatocyte plasma membrane bears receptors for the circumsporozoite protein of Plasmodium falciparum sporozoites. Cell. 1992 Sep 18;70(6):1021-33. doi: 10.1016/0092-8674(92)90251-7. PMID 1326407
- [Background] CDC (2020) 'CDC - Malaria - Malaria Worldwide - Impact of Malaria'. Available in: https://www.cdc.gov/malaria/malaria_worldwide/impact.html
- [Background] Clyde DF. Immunization of man against falciparum and vivax malaria by use of attenuated sporozoites. Am J Trop Med Hyg. 1975 May;24(3):397-401. doi: 10.4269/ajtmh.1975.24.397. PMID 808142
- [Background] Clyde DF, McCarthy VC, Miller RM, Hornick RB. Specificity of protection of man immunized against sporozoite-induced falciparum malaria. Am J Med Sci. 1973 Dec;266(6):398-403. doi: 10.1097/00000441-197312000-00001. No abstract available. PMID 4590095
- [Background] Cochrane AH, Aikawa M, Jeng M, Nussenzweig RS. Antibody-induced ultrastructural changes of malarial sporozoites. J Immunol. 1976 Mar;116(3):859-67. PMID 815435
- [Background] Cochrane AH, Nardin EH, de Arruda M, Maracic M, Clavijo P, Collins WE, Nussenzweig RS. Widespread reactivity of human sera with a variant repeat of the circumsporozoite protein of Plasmodium vivax. Am J Trop Med Hyg. 1990 Nov;43(5):446-51. doi: 10.4269/ajtmh.1990.43.446. PMID 2122747
- [Background] Collins WE, Jeffery GM. A retrospective examination of sporozoite- and trophozoite-induced infections with Plasmodium falciparum in patients previously infected with heterologous species of Plasmodium: effect on development of parasitologic and clinical immunity. Am J Trop Med Hyg. 1999 Jul;61(1 Suppl):36-43. doi: 10.4269/tropmed.1999.61-036. PMID 10432043
- [Background] Collins WE, Sullivan JS, Morris CL, Galland GG, Richardson BB. Observations on the biological nature of Plasmodium vivax sporozoites. J Parasitol. 1996 Apr;82(2):216-9. PMID 8604086
- [Background] Comer RD, Young MD, Porter JA Jr, Gauld JR, Merritt W. Chloroquine resistance in Plasmodium falciparum malaria on the Pacific coast of Colombia. Am J Trop Med Hyg. 1968 Nov;17(6):795-9. doi: 10.4269/ajtmh.1968.17.795. No abstract available. PMID 4881949
- [Background] Charoenvit Y, Collins WE, Jones TR, Millet P, Yuan L, Campbell GH, Beaudoin RL, Broderson JR, Hoffman SL. Inability of malaria vaccine to induce antibodies to a protective epitope within its sequence. Science. 1991 Feb 8;251(4994):668-71. doi: 10.1126/science.1704150.
- [Background] Chitnis CE. Molecular insights into receptors used by malaria parasites for erythrocyte invasion. Curr Opin Hematol. 2001 Mar;8(2):85-91. doi: 10.1097/00062752-200103000-00005. PMID 11224682
- [Result] Arevalo-Herrera M, Vera O, Castellanos A, Cespedes N, Soto L, Corradin G, Herrera S. Preclinical vaccine study of Plasmodium vivax circumsporozoite protein derived-synthetic polypeptides formulated in montanide ISA 720 and montanide ISA 51 adjuvants. Am J Trop Med Hyg. 2011 Feb;84(2 Suppl):21-7. doi: 10.4269/ajtmh.2011.10-0110. PMID 21292874